CLINICAL TRIAL: NCT06633276
Title: Nanopore Sequencing for Accelerating Breast Cancer Diagnosis in Tanzania: A Prospective Observational Study
Brief Title: Fast and Accurate Breast Cancer Diagnosis Using Nanopore Sequencing in Tanzania (Fast-ABCD Sequencing)
Status: Recruiting | Type: Observational
Sponsor: University of Bonn (Other)
Collaborators: German Cancer Research Center (Other); Kilimanjaro Christian Medical Centre,Moshi,Tanzania (Unknown)
Responsible Party: Principal Investigator, Oliver Henke, Head of Working Group Global Oncology, Section Global Health, University Hospital Bonn, University of Bonn
Other Study IDs: 23Ac03011
Record Dates: First submitted 2024-10-01; First posted 2024-10-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Invasive
Keywords: Nanopore sequencing; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Excess tissue from SoC diagnosis of suspected invasive breast cancer is preserved for DNA extraction using commercial spin column kits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nanopore sequencing: All adult patients at with suspected diagnosis of breast cancer undergoing biopsy or surgical resection will be offered to participate in the study. After informed written consent excess tissue is preserved for DNA extraction using commercial spin column kits and will be further analyzed.

SUMMARY:
This pilot study will test the feasibility of using nanopore sequencing for breast cancer diagnosis in Tanzania. It aims to show that nanopore sequencing is non-inferior to the current standard of care, with the potential for faster and more cost-efficient results. By enhancing the speed and accuracy of diagnosis, this approach could improve treatment planning and outcomes for patients in resource-limited settings.

DETAILED DESCRIPTION:
Excess fresh tissue samples from patients with suspected breast cancer will undergo nanopore sequencing alongside the current standard of care (SoC), which includes histopathology and biomarker analysis for estrogen receptor, progesterone receptor, and human epidermal growth factor receptor 2 (HER2) status.

Low-pass whole genome sequencing and DNA methylation-based classification will potentially enable the diagnosis of invasive ductal breast cancer in a cost-efficient and highly accurate manner. Additionally, breast cancer subtypes can be determined using methylation signatures and HER2 focal amplification, with results available within hours in a point-of-care setting.

The primary outcome measures are non-inferiority compared to SoC, turnaround time, and overall feasibility. Treatment is not altered due to results of the nanopore sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected diagnosis of breast cancer undergoing biopsy or surgical resection after specialist consultation as per institutional guidelines
* Excess fresh tumor sample
* Written informed consent

Exclusion Criteria:

* Unable to provide informed consent
* Patients who have already commenced therapy for BC (except for treatment other than biomedicine, e.g. herbal medicines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected invasive breast cancer undergoing diagnostic workup will be offered to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of nanopore-based biomarker evaluation | Concordance will be assessed after the enrollment of each cohort of 25 patients, with the final evaluation after study completion, approximately 12 months from enrollment start.
  Concordance of invasive breast cancer diagnosis using nanopore sequencing vs. IHC HR/HER2 status as standard of care. The concordance will be expressed as the percentage agreement between the two methods across 100 patients.
Feasibility | The ratio will be assessed continuously after the sequencing of each batch of samples, with the final evaluation at study completion, approximately 12 months from enrollment start.
  Feasibility will be measured by calculating the ratio of samples that are successfully sequenced and analyzed using nanopore sequencing technology, compared to the total number of samples processed.
Turnaround time | Through study completion, an average of 1 year
  Turnaround time will be measured as the time (in days) from biopsy to the availability of the nanopore sequencing report, compared to the time from biopsy to the finalized pathology report.

SECONDARY OUTCOMES:
Quality of Life (QoL) as assessed by the EORTC-QLQ BR-45 questionnaire | Administered at baseline, 6 months and 12 months.
  Quality of Life (QoL) will be measured using the EORTC-QLQ BR-45 questionnaire. The questionnaire will be administered at baseline and at multiple time points during the study, with changes in QoL scores compared over time. It is available in Swahali and in case of illiteracy will be read to the patient.
Patient Reported Experiences (PREs) with diagnostic procedures using a custom questionnaire | Administered within 24-48 hours post-biopsy.
  Patient-reported experiences related to the diagnostic procedures, including the ease of sample collection, the perceived length of time for results, and overall comfort during procedures, will be assessed using a custom questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Henke, MD, Principal Investigator — Section Global Health, University Hospital Bonn
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided